CLINICAL TRIAL: NCT07208318
Title: Rescuing Visual Perception in Aging Adults by Restructuring the Alpha-Gamma Neural Code
Brief Title: Restructuring the Alpha-Gamma Code in Aging Vision
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Robert Reinhart, Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 4230E_2
Record Dates: First submitted 2025-09-15; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Aging; Visual Perception; Noninvasive Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- active stimulation (Experimental)
  Interventions: Device: High definition transcranial electrical current stimulation
- sham stimulation (Sham Comparator)
  Interventions: Device: High definition transcranial electrical current stimulation

INTERVENTIONS:
Device: High definition transcranial electrical current stimulation — Low-intensity and safe, noninvasive application of electrical current to the human scalp with the goal of gradually modulating levels of neuronal excitability.

SUMMARY:
Tests whether age-related visual deficits arise from disrupted alpha-gamma coupling in visual cortex (V1) and MT. Uses fMRI, source-resolved HD-EEG, and personalized complex-waveform HD-tACS to (1) quantify aging effects on phase-amplitude coupling, (2) drive PAC into a preferred "gamma-at-alpha-troughs" state, and (3) bidirectionally change perception by aligning gamma to alpha troughs vs peaks. Two five-day, double-blind, sham-controlled studies (n=120 each) target contrast sensitivity (V1) and 3D shape-from-motion (MT), aiming for mechanistic insight and remediation in older adults with implications for ADRD.

DETAILED DESCRIPTION:
The project probes a causal account of age-related perceptual decline by focusing on alpha-gamma phase-amplitude coupling (PAC) in early visual cortex and area MT. The central hypothesis is that aging alters both the magnitude and phase structure of alpha-gamma interactions, degrading visual performance; restoring a preferred configuration-gamma power nested at alpha troughs-should improve perception.

Multimodal methods combine structural/functional MRI, high-density EEG with source reconstruction, and individualized complex-waveform HD-tACS tuned to each participant's neuroanatomy and oscillatory frequencies. Three questions drive the work: (i) Do age-related deficits track changes in alpha-gamma PAC magnitude/phase? (ii) Can frequency-coupled HD-tACS enforce the preferred PAC configuration and enhance perception, especially in more impaired older adults? (iii) Is perception bidirectionally controllable by placing gamma at alpha troughs (facilitation) versus peaks (disruption)?

Two specific aims implement matched, five-day, within-subjects, double-blind, sham-controlled experiments with 120 participants each. Aim 1 targets early visual cortex to test whether contrast sensitivity deficits scale with age, spatial frequency, and noise, and whether personalized HD-tACS can optimize PAC to improve contrast perception. Aim 2 targets MT to test whether 3D shape-from-motion (parallax) judgments decline with age as a function of surface-point lifetime and simulated depth, and whether trough- versus peak-aligned stimulation can restructure PAC to enhance motion-based shape perception. Outcomes will establish mechanistic links between PAC and visual aging and evaluate a noninvasive, personalized intervention path relevant to age-related decline and ADRD.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age or older
* normal or corrected-to-normal visual acuity, color vision, and stereo vision

Exclusion Criteria:

* not pregnant,
* no metal implants in head,
* no implanted electronic devices,
* no history of neurological problems or head injury,
* no skin sensitivity,
* no claustrophobia,
* no dementia (normal Mini Mental State Examination between 24-30; Montreal Cognitive Assessment > 25)
* no depression (normal Beck Depression Inventory II <13; Geriatric Depression Scale < 10)
* no ophthalmological diseases (e.g., strabismus, glaucoma, cataract, macular degeneration)
* no history of psychosis
* no cognitive deficits (MMSE score>24; MoCA>25)
* cannot be taking any psychoactive medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2030-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
contrast sensitivity | Baseline (pre-stimulation) and immediately post-stimulation, collected on each of the 5 study days.
  Orientation identification task
3D structural-from-motion | Baseline (pre-stimulation) and immediately post-stimulation, collected on each of the 5 study days.
  surface point lifetime (unlimited, 12 and 2 successive views) on 3D discrimination task
phase-amplitude coupling | Baseline (pre-stimulation) and immediately post-stimulation, collected on each of the 5 study days.
  alpha phase, gamma amplitude coupling (magnitude of coherency)

IPD SHARING:
Plan to Share IPD: No